CLINICAL TRIAL: NCT06092099
Title: A Clinical Investigation to Collect Real-life Measurement Data to Allow Development of Mathematical Algorithms for the Updated TENA SmartCare Change Indicator.
Brief Title: Collecting Real-life Data for the Updated TENA SmartCare Change Indicator.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Essity Hygiene and Health AB (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: GASOLINA
Record Dates: First submitted 2023-10-13; First posted 2023-10-23 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Urinary Incontinence
MeSH Terms: conditions — Urinary Incontinence

STUDY DESIGN:
Intervention Model Description: All subjects in the study will use the device
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): Subjects wear the sensor part of the Change indicator system during a 15-day period.
  Interventions: Device: TENA SmartCare Change Indicator

INTERVENTIONS:
Device: TENA SmartCare Change Indicator — The TENA SmartCare Change Indicator is an accessory to absorbent incontinence products, intended for use on individual(s) with urinary incontinence who are dependent on one or more caregivers to change the absorbent incontinence product. The TENA SmartCare Change Indicator estimates the degree of urine saturation in the absorbent incontinence product and notifies the caregivers. This facilitates the caregiver's decision regarding when to change the absorbent incontinence product. As the current study is needed to validate the updated device, the full system will not be used, only the sensor part.

SUMMARY:
This study is an explorative, open, single-arm clinical investigation to collect real-life measurement data in order to assess the mathematical algorithms involved in TENA SmartCare Change Indicator.

DETAILED DESCRIPTION:
The purpose of this exploratory clinical investigation is to evaluate safety and to collect real-life measurement data using the updated TENA SmartCare Change Indicator. The collected data will be used to assess and develop the device related algorithms. These algorithms have been tested in a laboratory setting but real-life measurement data are to be collected to the aid in further product development.

ELIGIBILITY:
Inclusion Criteria:

* Be willing and able to provide informed consent to participate or, if unable to provide such consent, have a legal representative who is willing and able to provide informed consent on behalf of the resident.
* Be 18 years of age of older.
* Be cared for at the investigation site.
* Suffer from urinary incontinence.
* Be current user of TENA Slip, Flex, Pants or Comfort incontinence products or during the course of the study be willing to become user of TENA Slip Flex, Pants or Comfort incontinence products.
* If applicable, be on a stable regimen of medications for urinary incontinence.

Exclusion Criteria:

* Have frequent (daily) faecal incontinence in the pad or having severe problems with faecal incontinence as determined by the investigator.
* Have severe incontinence product related skin problems, as defined by the GLOBIAD categorization 2B (skin loss & infection).
* Have any type of indwelling or external urinary catheter(s).
* Be anuric.
* Be of childbearing potential as determined by the investigator.
* Be managed using another automated or digital health technology incontinence management device.
* Have responsive behaviors of sufficient severity, in the opinion of the care staff, to make participation impractical.
* Have any other condition that makes participation in the clinical investigation
* Have a life expectancy of less than 90 days or be in receipt of palliative/terminal care.
* Have participated in an investigational study of a drug, biologic, or device within 30 days prior to entering the clinical investigation or planned during the clinical investigation.
* Be dependent on either alcohol or recreational drugs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2023-11-02 (Actual); Primary Completion 2023-12-21 (Actual); Study Completion 2024-02-28 (Actual)

PRIMARY OUTCOMES:
Urine weight | 15 days
  Absorbing hygiene products used by the subjects are collected in the investigation and the urine weight is determined. The urine weight is then matched with the data measured by the sensor to obtain connect sensor raw data with a specific urine content of an absorbing hygiene products

SECONDARY OUTCOMES:
Number of safety related events | 15 days
  Reported adverse events and device deficiencies are collected during the study.
Caregiver assessment on urine saturation | 15 days
  At the collection of the used absorbing hygiene products the caregiver assess the urine content of the product. This is done by indicating on a 3-point scale if the product change was 1. early, 2. in time or 3. late.
Caregiver usability for sensor | 15 days
  Using a questionnaire at the end of the study data on the caregivers user experience with the sensor is collected using a 5-grade Likert scale were 1 is minimum and 5 maximum and 5 represents the better outcome.
Resident satisfaction with sensor | 15 days
  Using a questionnaire at the end of the study data on the residents satisfaction with the sensor is collected using a 5-grade Likert scale were 1 is minimum and 5 maximum and 5 represents the better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Roland Frösing, MD, Principal Investigator — VIP Hälsan Väst
Locations (1):
- Tre Stiftelser Änggårdsbacken, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: No